CLINICAL TRIAL: NCT00792454
Title: Reduction of Mortality Prior to and During the First 90 Days of Dialysis Through a Renal Rehabilitation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Responsible Party: Principal Investigator, James C Wasserman, principal investigator, MaineHealth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3399
Record Dates: First submitted 2008-11-14; First posted 2008-11-18 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Chronic Kidney Disease; End Stage Kidney Disease; Cardiovascular Disease
Keywords: Chronic kidney disease; End stage renal disease; Exercise; Cardiovascular disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Cardiovascular Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise training/renal rehabilitation (Experimental): Experimental arm will undergo 12 weeks of training in exercise, meditation, and nutrition education.
  Interventions: Behavioral: exercise training
- control (No Intervention): Control co-hort will receive usual chronic kidney disease care and no exercise, meditation or dietary education intervention.

INTERVENTIONS:
Behavioral: exercise training — Subjects will undergo renal rehabilitation in the form of guided exercises 2 times per week for 3 months. Subjects will be encouraged to walk for 1 hour on their own a third day of the week.Subjects will receive recommendations for cardiovascular, weight training and stretching exercises.
  Cardiovascular and strength capabilities of all subjects will be evaluated at the initial session in order to prescribe the appropriate exercise regimen. An exercise physiologist will conduct these evaluations using the Perceived Level of Exertion Subjects will also receive education and practice in mindful meditation and a heart healthy diet.
  Subjects will be encouraged to continue exercises, meditation, and healthy eating habits after the 3-month in-center program. Subjects will receive follow-up phone calls at 3-month intervals to encourage ongoing exercise, meditation, and healthy diet.
  Arms: exercise training/renal rehabilitation

SUMMARY:
The mortality rate of treated patients with end stage renal disease(ESRD)is 22 deaths patient-years at risk in 2006. Incident patients with ESRD are most vulnerable within the first 90 days of dialysis, with an annualized mortality rate of 50 deaths/100 patient years. The vast majority of these deaths are due to cardiovascular causes. As cardiac rehabilitation programs have shown a 20% reduction in one year overall mortality rate post myocardial infarction the investigator proposes that a similar type of rehabilitation program will also have a benificial effect on morbidity and mortality in patients with chronic kidney disease(CKD)and ESRD.The overall goal of this project is to study whether a renal rehabilitation program based on guided exercise implemented in patients with stage III and stage IV CKD can influence the mortality rate of these patients prior to and during the first 90 days of dialysis

Hypothesis:The application of a guided exercise program (renal rehabilitation) instituted in patients with stage III or Stage IV CKD will decrease the mortality rate prior to the initiation of renal replacement therapy.

Hypothesis:The application of renal rehabilitation during the late stages of CKD will decrease the mortality risk during the first 90 days of renal rehabilitation therapy.

Hypothesis:A guided exercise program will have an immediate and prolonged effect on activity levels, mental health and adaption to chronic illness in patients with advanced CKD.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 yo
* stage III CKD (GFR<60ml/min)
* stage IV CKD (GFR<30ml/min)

Exclusion Criteria:

* active angina pectoris
* lower extremity amputation with no prosthesis
* orthopedic disorder severly exacerbated by activity
* chronic lung disease resulting in significant shortness of breath or oxygen de-saturation at rest
* cerebro cascular disease manifested by ongoing TIAs
* malignant carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2008-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Mortality prior to and During the First 90 Days of Dialysis | 5 years

SECONDARY OUTCOMES:
Measurement of physical fitness and quality of life | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Maine Nephrology Associates, Portland, Maine, United States